CLINICAL TRIAL: NCT05688319
Title: Effect of Problem-Solving Training for Mothers With Special Needs Children: A Randomized Controlled Study
Brief Title: Effect of Problem-Solving Training
Acronym: AtaturkU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: Phd Nurgül Karakurt (Unknown)
Responsible Party: Principal Investigator, Kübra Gökalp, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2022/64
Record Dates: First submitted 2023-01-05; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Child Development Disorders, Pervasive; Problems Psychosocial; Mother-Infant Interaction
Keywords: Mothers; Problems Psychosocial
MeSH Terms: conditions — Child Development Disorders, Pervasive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The participants in the experimental group were divided into five groups of eight participants each according to the number of days they visited the center. The training was conducted face to face in the meeting room of the special education and rehabilitation center. Within the scope of the study, problem-solving training was conducted for the mothers in the experimental group in the study once a week for 10 weeks . The duration of each training session was 60-90 minutes. The weekly training sessions for all the experimental groups were completed on the same day.
  Interventions: Behavioral: Problem-Solving Training
- control group (No Intervention): The control group did not receive any training, and there was no interaction between the experimental group and the control group during the training period.

INTERVENTIONS:
Behavioral: Problem-Solving Training — Within the scope of the study, problem-solving training was conducted for the mothers in the experimental group in the study once a week for 10 weeks. The duration of each training session was 60-90 minutes.
  Arms: experimental group

SUMMARY:
The aim of this study, therefore, is to determine the effect of problem-solving training on the interpersonal problem-solving skills of mothers with special needs children. This study was a parallel randomized controlled trial. The mothers were sorted into control and experimental groups (40 experimental and 40 control groups). A personal information form and the Interpersonal Problem Solving Inventory (IPSI) were used to collect data in this research. The participants in the experimental group gived to problem solving training program while the control group was not exposed to any intervention.The data in the control and experimental groups were homogeneously distributed. There was no significant difference in the pre-training test scores for any of the dimensions , but the post-training test scores were significantly higher in the experimental group than in the control group. Intragroup analysis with the Wilcoxon sign-rank test showed that there were significant differences between the pre-training and post-training test scores in the experimental group. Interpersonal problem-solving skills can be improved by providing problem-solving training to the mothers of children with special needs. Based on the findings of this study, it is recommended that psychiatric nurses provide training to protect and improve the well-being of children with special needs and their families.

DETAILED DESCRIPTION:
Design Data Collection Instruments A personal information form and the Interpersonal Problem Solving Inventory were used to collect data in this research.

Personal Information Form This form was prepared by the researcher, and consists of eight questions that cover the following information: mother's age, mother's education level, income level, family type, number of children, diagnosis of the child with special needs, age of the child with special needs, and gender of the child with special needs.

Problem-Solving Training Program The researchers prepared the content of the training program based on relevant published literature, and the training program has been verified by three experts. The training was conducted by a researcher who is an expert in the field of psychiatric nursing. Before the start of the training, the mothers in the experimental group were taken to the meeting room and were asked to answer a preliminary test. The day and time for the training, which was conducted at the center, were then scheduled. The participants in the experimental group were divided into five groups of eight participants each according to the number of days they visited the center. The training was conducted face to face in the meeting room of the special education and rehabilitation center. Within the scope of the study, problem-solving training was conducted for the mothers in the experimental group in the study once a week for 10 weeks. The duration of each training session was 60-90 minutes. The weekly training sessions for all the experimental groups were completed on the same day.

In the first session of the problem-solving training, the group members met each other, set the rules for the training sessions, and defined the purpose of the meeting. The second and third sessions covered problem orientation, general problem-solving approaches, and alternative solutions. In the fourth and fifth sessions, the importance of recognizing and expressing feelings in real life was discussed. Additionally, the problem-solving styles of the members were discussed, with a focus on whether they had an inattentive, impulsive problem-solving style. In the sixth and seventh sessions, the avoidant style of problem solving, which is a negative problem-solving style, was discussed. Further, participants were asked to reflect on their problem-solving style. In the eighth and nineth sessions, problem-solving dialogue in fictitious and real-life situations was discussed. The skills learned were reviewed through a question-and-answer format. The tenth (and last) session was a general evaluation.

The pre-training test was conducted on the same day in the experimental group and the control group. The control group did not receive any training, and there was no interaction between the experimental group and the control group during the training period. When the training was completed in the experimental group, the post-training test was conducted in both groups of participants on the same day at the center.

ELIGIBILITY:
Inclusion Criteria:

* Having a child with special needs
* Being over the age of 18 years

Exclusion Criteria:

• Hearing and speech problems in the mother.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Interpersonal Problem Solving Inventory | 12 week
  The inventory was developed by Çam and Tümkaya to measure the interpersonal problem-solving approaches and skills of university students between the ages of 18 and 30 years. The lowest score that can be obtained from the scale is 50 and the highest score is 250. The high score obtained for each subscale indicates that the trait related to interpersonal problem solving is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No